CLINICAL TRIAL: NCT01155674
Title: Innate Immune Functions of Immature Neutrophils
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Professor Jérôme Pugin, University Hospitals of Geneva
Other Study IDs: CER 09-311
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-02

CONDITIONS: Sepsis; SIRS
Keywords: Innate immunity; Neutrophils; Band forms
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No samples retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sepsis patients: Patients presenting sepsis
- SIRS patients: Patients presenting with the systemic inflammatory response syndrome
- Healthy subjects: Healthy blood donors

SUMMARY:
Polymorphonuclear neutrophils, or granulocytes, are essential effector cells of the innate immune system against bacterial infections. Their role in sepsis has been long established as the primary phagocyte to clear the infectious process. In the early phase of sepsis, one observes a massive recruitment of immature neutrophils from the bone marrow into peripheral blood, the so-called "band forms" or "left shift cells". Despite the daily clinical use of neutrophil band forms count in the care of septic patients and their abundance in septic blood, no information exists on the fate of these cells, nor on their capacity to mount an efficient innate immune response. It is the goal of this proposal to study the fate and the innate immune functions of immature neutrophils obtained in patients with early septic shock. Immature neutrophils will be separated from mature neutrophils. The following functions will be studied ex vivo in mature vs. immature neutrophils from a series of patients with severe sepsis and septic shock: (1) surface expression of receptors of the innate immunity; (2) production of inflammatory mediators and reactive oxygen species in response to bacterial agonists; (3) chemotaxis; (4) phagocytosis of Gram-positive and Gram-negative bacteria; and (5) ex vivo viability (life span) and resistance to apoptosis. Importantly, the investigators have developed and mastered all in vitro assays and cell separation techniques necessary to address and answer these important questions. This project will undoubtedly shed light on the fate and function of a prominent leukocyte population circulating in patients with severe bacterial infections and sepsis.

DETAILED DESCRIPTION:
Objectives

1. Primary objective: To determine the innate immune functions of immature neutrophils in comparison to those from mature neutrophils, sampled from patients with severe sepsis and sepsis shock and in control patients (trauma patients and healthy donors (only mature neutrophils in the latter case)
2. Secondary objectives: To determine the fate and span life of immature neutrophils in comparison to mature neutrophils, sampled from patients with severe sepsis and sepsis shock and in control patients (trauma patients and healthy donors (only mature neutrophils in the latter case).

Inclusion criteria

* Patients with severe sepsis or septic shock (according to ACCP/FCCM standard definitions) with > 5% immature neutrophils.
* Patients with a noninfectious systemic inflammatory response syndrome (SIRS), e.g. patients with head trauma or multiple trauma with > 5% immature neutrophils.
* Healthy donors

Exclusion criteria

* Severe immunosuppression (e.g. HIV with < 200 CD4/mm3), treatment with glucocorticoids (> 300 mg hydrocortisone/day) or other immunosuppressive therapy
* Neutropenia (neutrophils < 0.5 G/l).
* Recent chemotherapy or administration of intravenous immunoglobulins within the last 4 weeks.

Endpoints

* Surface expression of receptors of the innate immunity in immature vs. mature neutrophils.
* Production by immature vs. mature neutrophils of inflammatory mediators and reactive oxygen species in response to bacterial agonists.
* Chemotaxis of immature vs. mature neutrophils.
* Phagocytosis of Gram-positive and Gram-negative bacteria by immature vs. mature neutrophils.
* Ex vivo viability and resistance to apoptosis of immature vs. mature neutrophils.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis or septic shock (according to ACCP/FCCM standard definitions) with > 5% immature neutrophils.
* Patients with a noninfectious systemic inflammatory response syndrome (SIRS), e.g. patients with head trauma or multiple trauma with > 5% immature neutrophils.
* Healthy donors

Exclusion Criteria:

* Severe immunosuppression (e.g. HIV with < 200 CD4/mm3), treatment with glucocorticoids (> 300 mg hydrocortisone/day) or other immunosuppressive therapy
* Neutropenia (neutrophils < 0.5 G/l).
* Recent chemotherapy or administration of intravenous immunoglobulins within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with severe sepsis or septic shock
  * Patients with a noninfectious systemic inflammatory response syndrome (SIRS)
  * Healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Innate immune functions of neutrophils | 12 months
  * Surface expression of receptors of the innate immunity in immature vs. mature neutrophils.
  * Production by immature vs. mature neutrophils of inflammatory mediators and reactive oxygen species in response to bacterial agonists.
  * Chemotaxis of immature vs. mature neutrophils.
  * Phagocytosis of Gram-positive and Gram-negative bacteria by immature vs. mature neutrophils.
  * Ex vivo viability and resistance to apoptosis of immature vs. mature neutrophils.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Intensive Care, Geneva, Switzerland